CLINICAL TRIAL: NCT03278756
Title: Online Cognitive Control Training for Remitted Depressed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B/14730/RMD
Record Dates: First submitted 2017-08-18; First posted 2017-09-12 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Major Depression in Remission
Keywords: Depression; Remission; Relapse prevention; Cognitive control training; Internet intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Between subjects-design with two training conditions. The training condition is the only difference between the two groups during the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Control Training (Experimental): A cognitive control training, consisting of 10 sessions of 15 minutes each, will be administered. The task in this training is an adaptive paced auditory serial addition task, where participants need to click on the sum of the last two heard digits.
  Interventions: Behavioral: Cognitive control training
- Active Control Training (Active Comparator): An active control training, consisting of 10 sessions of 15 minutes each, will be administered. The task in this training is an adaptive low load cognitive task, where participants need to click on the last heard digit.
  Interventions: Behavioral: Active control training

INTERVENTIONS:
Behavioral: Cognitive control training — 10 sessions of an adaptive paced auditory serial addition task, each lasting 15 minutes, over the course of two weeks.
  Arms: Cognitive Control Training
Behavioral: Active control training — 10 sessions of an low cognitive load task, each lasting 15 minutes, over the course of two weeks.
  Arms: Active Control Training

SUMMARY:
This study evaluates the effectiveness of an internet-delivered cognitive control training as a preventive intervention for remitted depressed patients. Half of the participants will receive a cognitive control training, while the other half will receive a low cognitive load training that acts as an active control condition.

DETAILED DESCRIPTION:
Prospective studies have linked impaired cognitive control to increased cognitive vulnerability for future depression. Importantly, experimental studies indicate that cognitive control training can be used to reduce rumination and depressive symptomatology in MDD (major depressive disorder) and RMD (remitted depressed) samples. Provided that remitted depressed patients form a high-risk group for developing future depressive episodes, the current study will explore whether an internet-delivered cognitive control training can be used to reduce vulnerability for future depression in remitted depressed patients.

A computer training, consisting of 10 sessions of 15 minutes each, will be administered to participants, which are remitted depressed patients. This training can either be a cognitive control training, using an adaptive paced auditory serial addition task, or an active control training, with a low cognitive load task.

Dependent variables will be assessed pre- and post-training, as well as 3 and 6 months after the training, and consist of depressive symptomatology, related variables and cognitive control measures.

ELIGIBILITY:
Inclusion Criteria:

* History of ≥ 1 depressive episodes (major or bipolar)
* Currently in stable full or partial remission (≥ 3 months)

Exclusion Criteria:

* Major depressive disorder (current or less than 3 months in remission)
* Bipolar disorder (current or less than 3 months in remission)
* Psychotic disorder (current and/or previous)
* Neurological impairments (current and/or previous)
* Excessive substance abuse (current and/or previous)
* No ongoing psychotherapeutic treatment (maintenance treatment is allowed, but with a frequency of less than once every three weeks)
* Use of antidepressant medication is allowed if kept at a constant level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptomatology | Assessed at pre-training assessment and at 6 months follow-up
  Measured by the Beck Depression Inventory - II (BDI-II)
Change in depressive symptomatology | Assessed at pre-training assessment, at post-training assessment (within 1 week of completing the training), at 3 months follow-up and at 6 months follow-up
  Measured by the Depression Anxiety Stress Scales (DASS)
Change in depressive rumination (brooding) | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the Ruminative Response Scale (RRS), especially the brooding subscale

SECONDARY OUTCOMES:
Change in cognitive emotion regulation strategies | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the Cognitive Emotion Regulation Questionnaire (CERQ)
Change in quality of life | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the Quality of Life in Depression Scale (QLDS)
Remission from depression | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the Remission of Depression Questionnaire (RDQ)
Resilience | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the Connor-Davidson Resilience Scale (CD-RISC)

OTHER OUTCOMES:
User engagement | Assessed at post-training assessment (within 1 week of completing the training) and at 3 months follow-up
  Measured by the User Engagement Scale (UES)
Threatening experiences | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the List of Threatening Experiences (LTE)
Effortful control | Assessed at pre-training assessment and at 6 months follow-up
  Measured by the subscale Effortful Control (EC) from the Adult Temperament Questionnaire (ATQ)
Credibility and Expectancy | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the Credibility/Expectancy Questionnaire
Behavioral measure for cognitive control | Assessed at pre- and post-training assessment (within 1 week of completing the training) and at 3 and 6 months follow-up
  Measured by the non-adaptive Paced Auditory Serial Addition Task (PASAT)

CONTACTS AND LOCATIONS:
Overall Officials: Ernst HW Koster, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided